CLINICAL TRIAL: NCT00321711
Title: A Randomized, Double Blind, Placebo Controlled Study Evaluating the Efficacy and Safety of Romiplostim (AMG 531) Treatment of Subjects With Low or Intermediate Risk Myelodysplastic Syndrome (MDS) Receiving Hypomethylating Agents
Brief Title: Determination of Safe and Effective Dose of Romiplostim (AMG 531) in Subjects With Myelodysplastic Syndrome (MDS)Receiving Hypomethylating Agents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20050232
Record Dates: First submitted 2006-05-02; First posted 2006-05-04 (Estimated); Results first posted 2011-04-05 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-09

CONDITIONS: MDS; Myelodysplastic Syndromes; Thrombocytopenia
Keywords: MDS; Myelodysplastic Syndromes; Refractory Cytopenias; Thrombocytopenia
MeSH Terms: conditions — Myelodysplastic Syndromes; Thrombocytopenia; Cytopenia | interventions — romiplostim; Azacitidine; Decitabine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- Dose level 1 500 AMG 531 (Part A - azacitidine) (Active Comparator): 500 mcg AMG 531 weekly via subcutaneous injection + 75 mg/m2 azacitidine for 4 cycles
  Interventions: Biological: AMG 531 (Romiplostim); Drug: Azacitidine
- Dose level 1 750 AMG 531 (Part B - decitabine) (Active Comparator): 750 mcg AMG 531 weekly via subcutaneous injection + 20 mg/m2 decitabine for 4 cycles
  Interventions: Biological: AMG 531 (Romiplostim); Drug: Decitabine
- Dose level 2 750 AMG 531 (Part A - azacitidine) (Active Comparator): 750 mcg AMG 531 weekly via subcutaneous injection + 75 mg/m2 azacitidine for 4 cycles
  Interventions: Biological: AMG 531 (Romiplostim); Drug: Azacitidine
- Placebo (Part A - azacitidine) (Placebo Comparator): Placebo weekly via subcutaneous injection + 75 mg/m2 azacitidine for 4 cycles
  Interventions: Drug: Placebo; Drug: Azacitidine
- Placebo (Part B - decitabine) (Placebo Comparator): Placebo weekly via subcutaneous injection + 20 mg/m2 decitabine for 4 cycles
  Interventions: Drug: Placebo; Drug: Decitabine

INTERVENTIONS:
Drug: Placebo — Subjects in the control group will receive a placebo subcutaneous injection on a weekly basis during the 4 cycle treatment period.
  Arms: Placebo (Part A - azacitidine); Placebo (Part B - decitabine)
Biological: AMG 531 (Romiplostim) — AMG 531 (Romiplostim) will be administered weekly by subcutaneous injection at a dose of 500 or 750 μg during Part A and 750 μg during Part B for the 4 cycle treatment period, depending on randomization.
  Arms: Dose level 1 500 AMG 531 (Part A - azacitidine); Dose level 1 750 AMG 531 (Part B - decitabine); Dose level 2 750 AMG 531 (Part A - azacitidine)
Drug: Azacitidine — hypomethylating agent
  Arms: Dose level 1 500 AMG 531 (Part A - azacitidine); Dose level 2 750 AMG 531 (Part A - azacitidine); Placebo (Part A - azacitidine)
Drug: Decitabine — hypomethylating agent
  Arms: Dose level 1 750 AMG 531 (Part B - decitabine); Placebo (Part B - decitabine)

SUMMARY:
The purpose of this study is to evaluate the effect of Romiplostim (AMG 531) on the incidence of clinically significant thrombocytopenic events (grade 3 or 4 and/or receipt of platelet transfusions) in subjects with low or intermediate risk Myelodysplastic Syndrome (MDS) receiving hypomethylating agents. It is hypothesized that Romiplostim administration, at the appropriate dose and schedule, will result in reduction in the incidence of clinically significant thrombocytopenic events in low or intermediate risk MDS subjects receiving hypomethylating agents.

ELIGIBILITY:
Inclusion Criteria: - Diagnosis of MDS by bone marrow biopsy based on the World Health Organization (WHO) classification - Low, Intermediate-1 or Intermediate-2 risk category MDS using the IPSS (International Prognostic Scoring System) - Planned to receive either azacytidine 75 mg/m2 by subcutaneous administration each day for 7 days or decitabine 20 mg/m2 by intravenous administration each day for 5 days for at least 4 cycles Exclusion Criteria:

* Prior exposure to >3 cycles hypomethylating agents
* Prior history of leukemia or aplastic anemia
* Prior history of bone marrow transplantation
* Prior malignancy (other than in situ cervical cancer or basal cell cancer of the skin) unless treated with curative intent and without evidence of disease for ³ 3 years before randomization
* Active or uncontrolled infections
* Unstable angina, congestive heart failure [NYHA (New York Heart Association) > class II], uncontrolled hypertension [diastolic > 100 mmHg], uncontrolled cardiac arrhythmia, or recent (within 1 year) myocardial infarction
* History of arterial thrombosis ( eg, stroke or transient ischemic attack) in the past year
* History of venous thrombosis that currently requires anti-coagulation therapy
* Received IL-11 within 4 weeks of screening
* Less than 4 weeks since receipt of any therapeutic drug or device that is not FDA approved for any indication
* Have previously received any other thrombopoietic growth factor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2006-10-01 (Actual); Primary Completion 2009-10-19 (Actual); Study Completion 2009-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Greenberg PL, Garcia-Manero G, Moore M, Damon L, Roboz G, Hu K, Yang AS, Franklin J. A randomized controlled trial of romiplostim in patients with low- or intermediate-risk myelodysplastic syndrome receiving decitabine. Leuk Lymphoma. 2013 Feb;54(2):321-8. doi: 10.3109/10428194.2012.713477. Epub 2012 Nov 15. PMID 22906162
- [Background] Kantarjian HM, Giles FJ, Greenberg PL, Paquette RL, Wang ES, Gabrilove JL, Garcia-Manero G, Hu K, Franklin JL, Berger DP. Phase 2 study of romiplostim in patients with low- or intermediate-risk myelodysplastic syndrome receiving azacitidine therapy. Blood. 2010 Oct 28;116(17):3163-70. doi: 10.1182/blood-2010-03-274753. Epub 2010 Jul 14. PMID 20631375
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants in Part A were enrolled from 9 November 2006 through 31 August 2007; participants in Part B were enrolled from 26 March 2008 through 3 November 2008. Participants who enrolled in Part A were not eligible for enrollment in Part B.
Groups:
- Romiplostim (AMG 531) Placebo Plus Azacitidine: Romiplostim (AMG 531) placebo weekly via subcutaneous injection plus 75 mg/m^2 azacitidine daily for 7 days during each of four 28-day cycles (Part A)
- Romiplostim (AMG 531) 500 mcg Plus Azacitidine: 500 mcg romiplostim (AMG 531) weekly via subcutaneous injection plus 75 mg/m^2 azacitidine daily for 7 days during each of four 28-day cycles (Part A)
- Romiplostim (AMG 531) 750 mcg Plus Azacitidine: 750 mcg romiplostim (AMG 531) weekly via subcutaneous injection plus 75 mg/m^2 azacitidine daily for 7 days during each of four 28-day cycles (Part A)
- Romiplostim (AMG 531) Placebo Plus Decitabine: Romiplostim (AMG 531) placebo weekly via subcutaneous injection plus 20 mg/m^2 decitabine daily for 5 days during each of four 28-day cycles (Part B)
- Romiplostim (AMG 531) 750 mcg Plus Decitabine: 750 mcg romiplostim (AMG 531) weekly via subcutaneous injection plus 20 mg/m^2 decitabine daily for 5 days during each of four 28-day cycles (Part B)
Period: Part A
Arm/Group | Romiplostim (AMG 531) Placebo Plus Azacitidine | Romiplostim (AMG 531) 500 mcg Plus Azacitidine | Romiplostim (AMG 531) 750 mcg Plus Azacitidine | Romiplostim (AMG 531) Placebo Plus Decitabine | Romiplostim (AMG 531) 750 mcg Plus Decitabine
Started | 13 | 13 | 14 | 0 | 0
Completed | 8 (Participants in Part A were not eligible for enrollment in Part B) | 3 (Participants in Part A were not eligible for enrollment in Part B) | 3 (Participants in Part A were not eligible for enrollment in Part B) | 0 | 0
Not Completed | 5 | 10 | 11 | 0 | 0
Not completed — Adverse Event | 3 | 3 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0 | 0
Not completed — Disease progression | 0 | 1 | 0 | 0 | 0
Not completed — Requirement for alternative therapy | 0 | 2 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 3 | 0 | 0
Not completed — Other | 1 | 2 | 3 | 0 | 0
Not completed — Protocol deviation | 0 | 0 | 1 | 0 | 0
Period: Part B
Arm/Group | Romiplostim (AMG 531) Placebo Plus Azacitidine | Romiplostim (AMG 531) 500 mcg Plus Azacitidine | Romiplostim (AMG 531) 750 mcg Plus Azacitidine | Romiplostim (AMG 531) Placebo Plus Decitabine | Romiplostim (AMG 531) 750 mcg Plus Decitabine
Started | 0 (Participants in Part A were not eligible for enrollment in Part B) | 0 (Participants in Part A were not eligible for enrollment in Part B) | 0 (Participants in Part A were not eligible for enrollment in Part B) | 14 | 15
Completed | 0 | 0 | 0 | 8 | 10
Not Completed | 0 | 0 | 0 | 6 | 5
Not completed — Noncompliance | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 1
Not completed — Disease progression | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 2
Not completed — Death | 0 | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Romiplostim (AMG 531) Placebo Plus Azacitidine | Romiplostim (AMG 531) 500 mcg Plus Azacitidine | Romiplostim (AMG 531) 750 mcg Plus Azacitidine | Romiplostim (AMG 531) Placebo Plus Decitabine | Romiplostim (AMG 531) 750 mcg Plus Decitabine | Total
Number analyzed (Participants) | 13 | 13 | 14 | 14 | 15 | 69
Age, Continuous [Mean (Full Range); unit: Years] | 67.3 [58 to 86] | 71.9 [56 to 86] | 71.4 [61 to 81] | 70.5 [52 to 84] | 68.2 [55 to 81] | 69.8 [52 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 7 | 3 | 7 | 26
  Male | 7 | 10 | 7 | 11 | 8 | 43
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Caucasian | 13 | 10 | 14 | 9 | 11 | 57
  Black or African American | 0 | 2 | 0 | 1 | 1 | 4
  Hispanic or Latino | 0 | 0 | 0 | 2 | 3 | 5
  Asian | 0 | 1 | 0 | 2 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of a Clinically Significant Thrombocytopenic Event
Description: Occurrence of a clinically significant thrombocytopenic event within the participant, defined as any platelet count obtained from day 15 of cycle 1 through the end of the interim follow-up visit that was less than 50 x 10^9/L or receipt of platelet transfusions at any time through the interim follow-up visit.
Time Frame: Treatment period (up to 20 weeks)
Population: Full Analysis Set, composed of all randomized participants
Measure: Number; unit: Participants
Arm/Group | Romiplostim (AMG 531) Placebo Plus Azacitidine | Romiplostim (AMG 531) 500 mcg Plus Azacitidine | Romiplostim (AMG 531) 750 mcg Plus Azacitidine | Romiplostim (AMG 531) Placebo Plus Decitabine | Romiplostim (AMG 531) 750 mcg Plus Decitabine
Number analyzed (Participants) | 13 | 13 | 14 | 14 | 15
Participants | 11 | 8 | 10 | 11 | 12
Statistical Analysis 1: Comparison: Romiplostim (AMG 531) Placebo Plus Decitabine vs Romiplostim (AMG 531) 750 mcg Plus Decitabine; Test type: Superiority or Other; Odds Ratio (OR) = 1.032, 95% CI [0.153 to 6.950]
Statistical Analysis 2: Comparison: Romiplostim (AMG 531) Placebo Plus Azacitidine vs Romiplostim (AMG 531) 750 mcg Plus Azacitidine; Test type: Superiority or Other; Odds Ratio (OR) = 0.333, 95% CI [0.028 to 3.926]
Statistical Analysis 3: Comparison: Romiplostim (AMG 531) Placebo Plus Azacitidine vs Romiplostim (AMG 531) 500 mcg Plus Azacitidine; Test type: Superiority or Other; Odds Ratio (OR) = 0.118, 95% CI [0.007 to 1.882] — Adjusted by the stratification factor

2. Secondary Outcome: Hypomethylating Agent Dose Reduction and Delay Due to Thrombocytopenia
Description: Occurrence of hypomethylating agent dose reduction and delay due to thrombocytopenia
Time Frame: Treatment period (up to 20 weeks)
Population: Full Analysis Set, composed of all randomized participants
Measure: Number; unit: Participants
Arm/Group | Romiplostim (AMG 531) Placebo Plus Azacitidine | Romiplostim (AMG 531) 500 mcg Plus Azacitidine | Romiplostim (AMG 531) 750 mcg Plus Azacitidine | Romiplostim (AMG 531) Placebo Plus Decitabine | Romiplostim (AMG 531) 750 mcg Plus Decitabine
Number analyzed (Participants) | 13 | 13 | 14 | 14 | 15
Participants | 1 | 1 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Romiplostim (AMG 531) Placebo Plus Azacitidine vs Romiplostim (AMG 531) 500 mcg Plus Azacitidine; Test type: Superiority or Other; Odds Ratio (OR) = 1.000, 95% CI [0.063 to 15.988] — Romiplostim/placebo

3. Secondary Outcome: Achieving an Overall Response (Complete or Partial Response, CR or PR) at the End of the Treatment Period
Description: CR = decrease in bone marrow blast (≤5%) and improvement in peripheral blood counts (Hgb ≥ 11 g/dL, platelets ≥ 100x10^9/L, neutrophils ≥ 1x10^9/L, peripheral blasts=0%). PR = improvement in peripheral blood counts plus a decrease in bone marrow blasts ≥50% but not ≤5, or decrease in International Prognostic Scoring System score.
Time Frame: Treatment period (up to 20 weeks)
Population: Full Analysis Set, composed of all randomized participants
Measure: Number; unit: Participants
Arm/Group | Romiplostim (AMG 531) Placebo Plus Azacitidine | Romiplostim (AMG 531) 500 mcg Plus Azacitidine | Romiplostim (AMG 531) 750 mcg Plus Azacitidine | Romiplostim (AMG 531) Placebo Plus Decitabine | Romiplostim (AMG 531) 750 mcg Plus Decitabine
Number analyzed (Participants) | 13 | 13 | 14 | 14 | 15
Participants | 2 | 1 | 1 | 3 | 5
Statistical Analysis 1: Comparison: Romiplostim (AMG 531) Placebo Plus Decitabine vs Romiplostim (AMG 531) 750 mcg Plus Decitabine; Test type: Superiority or Other; Odds Ratio (OR) = 1.827, 95% CI [0.347 to 9.618] — Romiplostim/placebo
Statistical Analysis 2: Comparison: Romiplostim (AMG 531) Placebo Plus Azacitidine vs Romiplostim (AMG 531) 750 mcg Plus Azacitidine; Test type: Superiority or Other; Odds Ratio (OR) = 0.445, 95% CI [0.037 to 5.325] — Romiplostim/placebo
Statistical Analysis 3: Comparison: Romiplostim (AMG 531) Placebo Plus Azacitidine vs Romiplostim (AMG 531) 500 mcg Plus Azacitidine; Test type: Superiority or Other; Odds Ratio (OR) = 0.444, 95% CI [0.032 to 6.080] — Romiplostim/placebo

4. Secondary Outcome: Platelet Transfusion
Description: Occurrence of one or more platelet transfusions from study day 1 through the interim follow-up visit (16 weeks)
Time Frame: Study day 1 through the interim follow-up visit (up to 20 weeks)
Population: Full Analysis Set, composed of all randomized participants
Measure: Number; unit: Participants
Arm/Group | Romiplostim (AMG 531) Placebo Plus Azacitidine | Romiplostim (AMG 531) 500 mcg Plus Azacitidine | Romiplostim (AMG 531) 750 mcg Plus Azacitidine | Romiplostim (AMG 531) Placebo Plus Decitabine | Romiplostim (AMG 531) 750 mcg Plus Decitabine
Number analyzed (Participants) | 13 | 13 | 14 | 14 | 15
Participants | 9 | 6 | 5 | 8 | 7
Statistical Analysis 1: Comparison: Romiplostim (AMG 531) Placebo Plus Azacitidine vs Romiplostim (AMG 531) 750 mcg Plus Azacitidine; Test type: Superiority or Other; Difference in incidence rate = -33.5, 95% CI [-69.0 to 2.0] — Romiplostim - placebo
Statistical Analysis 2: Comparison: Romiplostim (AMG 531) Placebo Plus Decitabine vs Romiplostim (AMG 531) 750 mcg Plus Decitabine; Test type: Superiority or Other; Odds Ratio (OR) = 0.315, 95% CI [0.029 to 3.412]
Statistical Analysis 3: Comparison: Romiplostim (AMG 531) Placebo Plus Azacitidine vs Romiplostim (AMG 531) 500 mcg Plus Azacitidine; Test type: Superiority or Other; Odds Ratio (OR) = 0.211, 95% CI [0.021 to 2.082]

ADVERSE EVENTS:
Time Frame: Up to 20 weeks
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Part A Placebo | Part A Romiplostim 500 µg | Part A Romiplostim 750 µg | Part B Placebo | Part B Romiplostim 750 µg
Serious Adverse Events (participants affected / at risk) | 9/13 | 4/13 | 10/14 | 8/14 | 8/15
Other Adverse Events (participants affected / at risk) | 11/13 | 13/13 | 14/14 | 14/14 | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A Placebo (N=13) | Part A Romiplostim 500 µg (N=13) | Part A Romiplostim 750 µg (N=14) | Part B Placebo (N=14) | Part B Romiplostim 750 µg (N=15)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 1 | 1 | 3 | 4
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Caecitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Inflammation (General disorders) | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 1 | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Implant site infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 2 | 2 | 2
Pneumonia fungal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 2 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A Placebo (N=13) | Part A Romiplostim 500 µg (N=13) | Part A Romiplostim 750 µg (N=14) | Part B Placebo (N=14) | Part B Romiplostim 750 µg (N=15)
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 2 | 4 | 2
Anaemia haemolytic autoimmune (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Bone marrow disorder (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 2 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 4 | 2 | 9 | 4
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 0 | 0 | 3 | 2
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 2 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Abnormal sensation in eye (Eye disorders) | 0 | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Anal pruritus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 5 | 7 | 7 | 5 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 4 | 6 | 5 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrointestinal oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1
Gingival erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1
Gingival swelling (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 6 | 4 | 6 | 6 | 5
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 0
Tongue discolouration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Tooth socket haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 1 | 1 | 2
Asthenia (General disorders) | 2 | 1 | 2 | 1 | 2
Catheter site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 1
Catheter site inflammation (General disorders) | 0 | 0 | 0 | 0 | 1
Catheter thrombosis (General disorders) | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 2 | 0 | 2
Cyst (General disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 5 | 4 | 2 | 3 | 2
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | 0
Infusion site haemorrhage (General disorders) | 0 | 1 | 0 | 0 | 0
Injection site discomfort (General disorders) | 0 | 0 | 2 | 0 | 0
Injection site erythema (General disorders) | 1 | 2 | 3 | 0 | 0
Injection site haematoma (General disorders) | 0 | 0 | 2 | 0 | 0
Injection site haemorrhage (General disorders) | 1 | 2 | 1 | 0 | 0
Injection site irritation (General disorders) | 1 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 2 | 2 | 4 | 0 | 0
Injection site pruritus (General disorders) | 1 | 1 | 1 | 0 | 0
Injection site rash (General disorders) | 0 | 2 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 1 | 2 | 0 | 0
Injection site swelling (General disorders) | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 4 | 2 | 2 | 3 | 3
Pain (General disorders) | 1 | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 1 | 0 | 3 | 4 | 3
Ulcer haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Hepatic cyst (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 2 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 3
Oral candidiasis (Infections and infestations) | 1 | 1 | 1 | 0 | 1
Oral fungal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Parotitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pharyngeal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 4 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 3 | 2 | 2 | 2
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood magnesium decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0 | 0
Cardiac murmur (Investigations) | 1 | 0 | 0 | 0 | 0
Heart sounds abnormal (Investigations) | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Pulmonary arterial pressure increased (Investigations) | 0 | 0 | 1 | 0 | 0
Reticulin increased (Investigations) | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 2 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3 | 5 | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 2 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Iron overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3 | 3 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Muscle swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 5 | 1 | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 4 | 3 | 2
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 1 | 1 | 2
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Mental impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Migraine with aura (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 0 | 2
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 2 | 1 | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 2 | 0 | 4 | 4
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Nervousness (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 2 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Penile discharge (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Scrotal erythema (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Scrotal swelling (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 1 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 1 | 1 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 1 | 3 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 3 | 0
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Blood blister (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 4 | 1 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 2 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 3 | 1 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Skin nodule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Vasculitic rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Breast lump removal (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 4 | 2 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Pallor (Vascular disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.